CLINICAL TRIAL: NCT01047267
Title: Pharmacokinetics of Anidulafungin in Critically Ill Patients With Invasive Candidiasis
Brief Title: Pharmacokinetics of Anidulafungin on Intensive Care Unit (ICU)
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JWC Alffenaar, PharmD, PhD, University Medical Center Groningen
Other Study IDs: ANIDULA-133
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Invasive Candidiasis; Critically Ill
Keywords: candidiasis; invasive fungal disease; critically ill; anidulafungin; pharmacokinetics
MeSH Terms: conditions — Candidiasis, Invasive; Critical Illness; Candidiasis; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to determine whether pharmacokinetic parameters of anidulafungin correlate with disease severity and plasma protein levels in critically ill patients.

DETAILED DESCRIPTION:
One of the risk factors for mortality of patients with candidemia is inadequate antifungal therapy. The first days in the intensive care unit (ICU), patients are unstable and it can be questioned whether therapeutic levels of anidulafungin are reached after a standard loading scheme. At this moment there are several clues that the PK of anidulafungin in critically ill patients is different, but an overall picture is lacking.

For the investigation of the correlation of the pharmacokinetics of anidulafungin and the disease severity a full pharmacokinetic profile will be obtained. Predictive scoring systems will be used to assess disease severity.

ELIGIBILITY:
Inclusion Criteria:

* treatment with anidulafungin
* at least 18 years of age
* invasive candidiasis
* admitted to an intensive care unit

Exclusion Criteria:

* allergic to anidulafungin or its excipients
* contra-indication stated in SPC
* neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with invasive candidiasis admitted to an intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To investigate the correlation of pharmacokinetic parameters of anidulafungin with markers for disease severity - either disease severity scores or parameters (singly, or combined) for inflammation or organ function - and plasma protein levels. | 3 days

SECONDARY OUTCOMES:
Time (in days) to culture conversion | max 28 days
Response to treatment at day 28 | 28 days
Mortality at day 28 due to fungal infection and overall mortality at 28 days | 28 days
AUC/MIC ratio, time above MIC | max 28 days
Composing a pharmacokinetic model of anidulafungin in critically ill patients | max 28 days

CONTACTS AND LOCATIONS:
Overall Officials: JWC Alffenaar, PharmD, PhD, Study Chair — University Medical Center Groningen; MJP van Wanrooy, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] van Wanrooy MJ, Proost JH, Rodgers MG, Zijlstra JG, Uges DR, Kosterink JG, van der Werf TS, Alffenaar JW. Limited-sampling strategies for anidulafungin in critically ill patients. Antimicrob Agents Chemother. 2015 Feb;59(2):1177-81. doi: 10.1128/AAC.03375-14. Epub 2014 Dec 8. PMID 25487797
- [Derived] van Wanrooy MJ, Rodgers MG, Uges DR, Arends JP, Zijlstra JG, van der Werf TS, Kosterink JG, Alffenaar JW. Low but sufficient anidulafungin exposure in critically ill patients. Antimicrob Agents Chemother. 2014;58(1):304-8. doi: 10.1128/AAC.01607-13. Epub 2013 Oct 28. PMID 24165173